CLINICAL TRIAL: NCT05179421
Title: A Dose Ranging Study for a Pharmacodynamic Model of Oxytocin for Peripheral Analgesia Effects
Brief Title: Dose Ranging Study of Intravenous Oxytocin for Analgesia to Heat Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00079629
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Each participant will receive 2 IV infusions separated by 1 hour One study day: saline (placebo) then oxytocin 1.3 micrograms Another study day: oxytocin 0.3 micrograms then oxytocin 7 micrograms
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- First infusion day low dose oxytocin, Second infusion day high dose oxytocin (Experimental): On the first oxytocin study day, participants will receive a 10 minute IV infusion of saline then one hour later will receive a 10 minute infusion of oxytocin 1.3 micrograms. On the second study day they will receive a 10 minute IV infusion of oxytocin 0.3 micrograms then one hour later will receive a 10 minute infusion of oxytocin 7 micrograms.
  Interventions: Drug: Low dose oxytocin; Drug: High dose oxytocin
- First infusion day high dose oxytocin, Second infusion day low dose oxytocin (Experimental): On the first oxytocin study day, participants will receive a 10 minute IV infusion of oxytocin 0.3 micrograms then one hour later will receive a 10 minute infusion of oxytocin 7 micrograms. On the second study day they will receive a 10 minute IV infusion of saline then one hour later will receive a 10 minute infusion of oxytocin 1.3 micrograms.
  Interventions: Drug: Low dose oxytocin; Drug: High dose oxytocin

INTERVENTIONS:
Drug: Low dose oxytocin — 10 minute IV infusion of saline followed by a 10 minute infusion of oxytocin 1.3 micrograms
  Other Names: Pitocin
Drug: High dose oxytocin — 10 minute IV infusion of oxytocin 0.3 micrograms followed by a 10 minute infusion of oxytocin 7 micrograms
  Other Names: Pitocin

SUMMARY:
This is a study of participants that will receive intravenous (IV) infusions of oxytocin (naturally occurring hormone that is made by the brain).

In this study healthy participants will be recruited for the study. There will be 3 study related visits: 1) screening and informed consent 2) study medication infusions and thermal heat testing 3) study medication infusions and thermal heat testing. During study visits 2 and 3 an IV catheter will be placed and a dose of oxytocin or placebo (inactive solution) will be given over a 10 minute period; 1 hour after the first infusion, a second 10 minute infusion of oxytocin will be administered.

Investigators will perform some tests to evaluate how oxytocin changes perceptions of the skin. Investigators will study a painful perception by placing a probe on the skin of the side of lower leg and heating it up to 113-117 degrees Fahrenheit (F) (45-47 degrees Celsius (C)) for 5 minutes. Each participant will score any pain that is experienced on a 0 to 10 scale for each minute during the heating period. Most people find that pain rises during the 5 minutes, but remains mild; usually less than 5 on the 0 to 10 pain scale. The temperature of the 5 minute heating will be determined according to the participants pain rating during the screening visit.

The primary objective of the study is to determine the dose response of IV oxytocin for analgesia (pain relief) to experimental heat pain.

DETAILED DESCRIPTION:
Equal numbers of adult men and women; ages 18-75 will be recruited. Participants will report to the research unit for three visits, 1) screening and informed consent 2) study medication infusions and thermal heat testing 3) study medication infusions and thermal heat testing separated by at least 72 hours.

For study infusion visits, study participants will come to the Clinical Research Unit and one intravenous (IV) catheter will be inserted in the forearm for oxytocin infusions. Participants in this study will receive a dose of oxytocin or placebo at a steady rate for 10 minutes; one hour later, a second dose of oxytocin will be administered during one visit. During the second study infusion visit, a lower dose of oxytocin will be given by a 10-minute IV infusion and one hour later a second infusion of oxytocin at a higher dose will be given. On one study day the doses will by 0 and 1.3 micrograms (µg) and on the other study day the doses will be 0.3 and 7 µg oxytocin. The order of study days will be randomized and double-blinded. As a result, each participant will receive oxytocin doses of 0, 0.3, 1.3, and 7 µg in this double blind design.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 and < 75 years of age, Body Mass Index (BMI) <40.
2. Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status 1, 2, or 3.
3. For healthy volunteers, normal blood pressure (systolic 90-140 mmHg; diastolic 50-90 mmHg) resting heart rate 45-100 beats per minute) without medication. For knee arthritis subjects, normal blood pressure or, for those with hypertension, pressure controlled with anti-hypertensives and with a resting heart rate 45-100 beats per minute.
4. Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full cycle before study drug administration.

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
2. Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
3. Women who are pregnant (positive result for serum pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years
4. Subjects with neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.
5. Subjects with current or history of ventricular tachycardia, atrial fibrillation or prolonged QT interval.
6. Subjects with past or current history of hyponatremia or at risk for hyponatremia; anyone taking thiazide diuretics, loop diuretics, combination diuretics, lithium, carbamazepine, enalapril, Ramipril, celecoxib, temazepam, gliclazide, glimepiride, glibenclamide, glipizide, omeprazole, pantoprazole, desmopressin, SSRI's, MAOI, or the recreational drug ecstasy.
7. Subjects with a known latex allergy.
8. Subjects with a pain score rating of 1 or less during the initial training session to a 5 minute heating of 45°C- 47 °C to the lower calf.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Infusion Day
Arm/Group | First Infusion Day Low Dose Oxytocin, Second Infusion Day High Dose Oxytocin | First Infusion Day High Dose Oxytocin, Second Infusion Day Low Dose Oxytocin
Started | 14 | 11
Completed | 13 | 11
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: At Least 5 Days Between Infusion Studies
Arm/Group | First Infusion Day Low Dose Oxytocin, Second Infusion Day High Dose Oxytocin | First Infusion Day High Dose Oxytocin, Second Infusion Day Low Dose Oxytocin
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0
Period: Second Infusion Day
Arm/Group | First Infusion Day Low Dose Oxytocin, Second Infusion Day High Dose Oxytocin | First Infusion Day High Dose Oxytocin, Second Infusion Day Low Dose Oxytocin
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: As noted in Participant Flow, there were 14 participants in Arm 1 and 11 participants in Arm 2. One subject in Arm 1 experienced near syncope during intravenous catheter insertion. This rapidly resolved spontaneously, but the subject did not further participate and did not receive study drug or undergo baseline testing.
Groups:
- Total: Total of all reporting groups
Arm/Group | First Infusion Day Low Dose Oxytocin, Second Infusion Day High Dose Oxytocin | First Infusion Day High Dose Oxytocin, Second Infusion Day Low Dose Oxytocin | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (14) | 42 (15) | 41 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 10 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Dose Response of Intravenous Oxytocin on Sustained Heat Pain
Description: Pain intensity was reported by the subject at the end of the 5 minute heating of the skin to 45 - 47 degrees C, using a verbal pain scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to THE WORST PAIN IMAGINABLE. Heating temperature was determined for each individual according to pain rating during screening visit. Pain scores obtained at 15, 30, and 45 minutes after the end of each 10 minute infusion were averaged for each individual and analyzed as th
Time Frame: 45 min after the end of each study drug infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: 10 minute intravenous infusion of saline placebo
- Oxytocin 0.3 mcg: 10 minute intravenous infusion of oxytocin, 0.3 mcg
- Oxytocin 1.3 mcg: 10 minute intravenous infusion of oxytocin, 1.3 mcg
- Oxytocin 7.0 mcg: 10 minute intravenous infusion of oxytocin, 7.0 mcg
Arm/Group | Placebo | Oxytocin 0.3 mcg | Oxytocin 1.3 mcg | Oxytocin 7.0 mcg
Number analyzed (Participants) | 24 | 24 | 24 | 24
units on a scale
  Prior to infusion | 3.1 (1.2) | 2.9 (1.1) | 3.1 (1.2) | 2.9 (1.1)
  15 minutes after end of infusion | 2.4 (1.5) | 2.4 (1.4) | 2.3 (1.3) | 2.3 (1.6)
  30 minutes after end of infusion | 2.5 (1.4) | 2.4 (1.4) | 2.3 (1.7) | 2.2 (1.3)
  45 minutes after end of infusion | 2.3 (1.5) | 2.3 (1.5) | 2.2 (1.5) | 2.1 (1.2)
  Average of 15, 30, and 45 min scores (Primary Outcome Measure) | 2.4 (1.4) | 2.4 (1.4) | 2.2 (1.4) | 2.2 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Oxytocin 0.3 mcg vs Oxytocin 1.3 mcg vs Oxytocin 7.0 mcg; Pain scores over time will first be modeled using NONMEM with derived parameters of maximum effect (Emax) and doses to produce a 50% and 90% maximum drug effect (C50 and C90, respectively), the steepness of the dose response curve (γ), and the time to peak effect. Inter-subject variability (e.g., biological variability) will evaluate additive, proportional, and exponential models. Residual intrasubject variability (e.g., noise) will typically require an additive and multiplicative error model; Test type: Other — NONMEM applies nonlinear mixed effects modeling to evaluate the relationship between predicted drug concentration after administration from known pharmacokinetics and a pharmacodynamic effect, in this case being a reduction in pain from sustained heat application; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: One week after each oxytocin infusion study day
Description: Peripheral oxyhemoglobin saturation, BP and HR will be measured non invasively before and 15, 30, and 60 min after each IV infusion. Participants were contacted daily for one week after each infusion study day and queried for any side effects.
Groups:
- Placebo Infusion: Ten minute intravenous infusion of placebo
- Oxytocin, 0.3 mcg Infusion: Ten minute intravenous infusion of oxytocin, 0.3 mcg
- Oxytocin, 1.3 mcg Infusion: Ten minute intravenous infusion of oxytocin, 1.3 mcg
- Oxytocin, 7.0 mcg Infusion: Ten minute intravenous infusion of oxytocin, 7.0 mcg
Arm/Group | Placebo Infusion | Oxytocin, 0.3 mcg Infusion | Oxytocin, 1.3 mcg Infusion | Oxytocin, 7.0 mcg Infusion
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
The original study design called for equal recruitment of subjects across three age ranges: young (18-39-year-old) middle (40 - 59-year-old) and older (60 - 75-year-old) with separate randomization in each group. The protocol was subsequently amended to remove this requirement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT05179421/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT05179421/ICF_000.pdf